CLINICAL TRIAL: NCT00865566
Title: Phase 2b, Randomized, Placebo-Controlled Test-of-Concept Trial to Evaluate the Safety and Efficacy of a Multiclade HIV-1 DNA Plasmid Vaccine Followed by a Multiclade HIV-1 Recombinant Adenoviral Vector Vaccine in HIV-Uninfected, Adenovirus Type 5 Neutralizing Antibody Negative, Circumcised Men and Male-to-Female (MTF) Transgender Persons, Who Have Sex With Men
Brief Title: Safety and Effectiveness of HIV-1 DNA Plasmid Vaccine and HIV-1 Recombinant Adenoviral Vector Vaccine in HIV-Uninfected, Circumcised Men and Male-to-Female (MTF) Transgender Persons Who Have Sex With Men
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was stopped for efficacy futility
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 505; 10753 (Registry Identifier: DAIDS ES); NCT00919789 (obsolete NCT alias)
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; HIV Treatment Vaccine; Adenovirus
MeSH Terms: conditions — HIV Infections; Adenoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive a recombinant DNA plasmid vaccine injection at study entry and on Days 28 and 56, followed by a recombinant adenoviral serotype vector vaccine injection on Day 168. As of April 2013, all vaccinations in this study have been stopped.
  Interventions: Biological: DNA plasmid vaccine; Biological: Recombinant adenoviral serotype 5 (rAD5) vector vaccine
- 2 (Placebo Comparator): Participants will receive a recombinant DNA plasmid vaccine placebo injection at study entry and on Days 28 and 56, followed by a recombinant adenoviral serotype vector vaccine placebo injection on Day 168. As of April 2013, all vaccinations in this study have been stopped.
  Interventions: Biological: DNA vaccine placebo; Biological: HIV-1 recombinant adenovirus vaccine placebo

INTERVENTIONS:
Biological: DNA plasmid vaccine — 4-mg injection administered as 1 mL intramuscularly (IM) via Biojector® in either deltoid
  Other Names: VRC-HIVDNA016-00-VP
  Arms: 1
Biological: Recombinant adenoviral serotype 5 (rAD5) vector vaccine — 1 x 10^10 particle units (PU) administered as 1mL IM by needle and syringe in either deltoid
  Other Names: VRC-HIVADV014-00-VP
  Arms: 1
Biological: DNA vaccine placebo — 1 mL IM via Biojector® in either deltoid
  Other Names: VRC-PBSPLA043-00-VP; phosphate buffered saline (PBS)
  Arms: 2
Biological: HIV-1 recombinant adenovirus vaccine placebo — 1 mL administered IM by needle and syringe in either deltoid
  Other Names: VRC-DILUENT013-DIL-VP; final formulation buffer (FFB)
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a VRC DNA/rAd5 vaccine regimen in healthy, circumcised men and male-to-female (MTF) transgender persons who have sex with men.

NOTES:

As of April 2013, all vaccinations in this study have been stopped.

As of June 2017, this study has been closed.

DETAILED DESCRIPTION:
In 2007, the Joint United Nations Programme on HIV/AIDS estimated that 33.2 million people were living with HIV/AIDS globally. The U.S. HIV prevalence data reported in October 2008 by the Centers for Disease Control and Prevention estimate that 1.1 million adults and adolescents were living with diagnosed or undiagnosed HIV infection in the United States at the end of 2006. Nearly half of all U.S. HIV infections (48.1%) were found in men who have sex with men (MSM). Given the difficulty of maintaining behaviors that prevent HIV transmission over a lifetime and the occurrence of nonconsensual sex, the need for a safe and effective vaccine is clear. The primary purpose of this study is to determine the safety and efficacy of a VRC DNA/rAd5 vaccine regimen in healthy, at-risk, circumcised men and MTF transgender persons who have sex with men.

Participants will be randomly assigned to one of two arms. Participants in Arm 1 will receive a recombinant DNA plasmid vaccine injection at study entry and on Days 28 and 56, followed by a recombinant adenoviral serotype vector vaccine injection on Day 168. Participants in Arm 2 will receive placebo injections at study entry and on Days 28, 56, and 168.

Participants who do not become HIV infected will be actively followed for a minimum of 24 months and will continue to be followed by the study for long-term safety surveillance for a total of 5 years following enrollment. Participants will be contacted annually during the period of long-term safety surveillance.

Participants who are found to be HIV infected prior to receiving their first injection or who receive their first injection but were HIV infected prior to study start will be followed on a modified schedule.

Participants who become HIV infected will be followed for 6 months post-diagnosis.

At most study visits, participants will undergo a physical exam and blood draw.

NOTES:

As of April 2013, all vaccinations in this study have been stopped. Participants have been notified of whether they received the study vaccines or placebo. Participants diagnosed with HIV infection will attend study visits for 6 months for health monitoring. Participants who are not diagnosed with HIV infection will attend planned study visits for 24 months and will be followed by the study clinic at least annually for a total of 5 years following study enrollment.

As of June 2017, this study has been closed. Therefore, to avoid further burden on study participants, further participant follow-up for the study is suspended.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 and -2 negative
* Good general health
* Fully circumcised
* Experienced one or both of the following HIV risk criteria in the 6 months before study entry:

  1. Unprotected anal intercourse with one or more male or MTF transgender partner(s)
  2. Anal intercourse with two or more male or MTF transgender partners
* Alanine aminotransferase (ALT) 2.5 or less times the upper limit of normal (ULN)
* Ad5 neutralizing antibody (nAb) titer less than 1:18
* Have access to a participating study site and are willing to be followed during the study
* Demonstrate understanding of the study
* Willing to receive HIV test results
* Willing to discuss HIV infection risks and amenable to risk-reduction counseling
* Agrees not to enroll in another study of an investigational research agent before unblinding of this study
* NOTE: MTF transgender volunteers who have undergone gender reassignment surgery (GRS) are eligible to participate if they provide documentation from a health care provider confirming that they were fully circumcised prior to GRS. MTF transgender volunteers who have not undergone GRS are eligible to participate if they meet all enrollment criteria. Receipt of hormonal therapy does not make a transgender volunteer ineligible.

Exclusion Criteria:

* HIV vaccines in prior HIV vaccine trial. Participants who can provide documentation that they received a placebo in a prior HIV trial may be eligible.
* Used antiretroviral (ARV) drugs for the purpose of HIV-1 prophylaxis for greater than or equal to 50% of days during the 3 months prior to first vaccination or for 30 consecutive days within the 60 days prior to first vaccination
* Circumcised within 90 days prior to first vaccination or displays evidence that surgical site is not fully healed
* Immunosuppressive medications within 168 days prior to first study vaccination. Participants who have used corticosteroid nasal sprays for allergic rhinitis; topical corticosteroids for mild, uncomplicated dermatitis; or oral/parenteral corticosteroids for nonchronic conditions are not excluded.
* Blood products within 90 days prior to first study vaccination
* Immunoglobulin within 90 days prior to first study vaccination
* Live attenuated vaccines other than influenza vaccine within 30 days prior to first study vaccination
* Investigational research agents within 90 days prior to first study vaccination
* Influenza vaccine or any vaccines that are not live attenuated within 14 days prior to first study vaccination
* Allergy treatment with antigen injections within 30 days prior to first study vaccination or that are scheduled within 14 days after first vaccination
* Clinically significant medical condition, physical examination findings, abnormal laboratory results, or past medical history that, in the judgment of the investigator, has significant implications for current health
* Any medical, psychiatric, or job-related responsibility that would interfere with the study. More information about this criterion can be found in the protocol.
* Any concern that, in the opinion of the investigator, may interfere with a participant's completion of the post-vaccination symptom log
* History of serious adverse reactions to vaccinations, including anaphylaxis or allergy to any of the vaccine's components
* Current anti-tuberculosis prophylaxis or therapy
* Autoimmune disease. People with mild, stable, and uncomplicated autoimmune disease that does not require immunosuppressive medication and that, in the judgment of the site investigator, is likely not subject to exacerbation and likely not to complicate reactogenicity and adverse event assessments are not excluded.
* Immunodeficiency
* Bleeding disorder
* History of malignancy
* Seizure disorder. People with a history of seizures who have had no seizures within the 3 years prior to study entry are not excluded.
* Asthma other than mild, well-controlled asthma
* Hereditary angioedema (HAE), acquired angioedema (AAE), or idiopathic angioedema

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2504 (Actual)
Dates: Start 2009-05; Primary Completion 2017-10-06 (Actual); Study Completion 2017-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Hammer, Study Chair — Columbia University; Magdalena Sobieszczyk, Study Chair — Columbia University; Michael Yin, Study Chair — Columbia University
Locations (22):
- United States (22):
  - Alabama CRS, Birmingham, Alabama
  - The AIDS Research Alliance of America CRS, Los Angeles, California
  - UCLA CARE Center CRS, Los Angeles, California
  - Bridge HIV CRS, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Orlando Immunology Center CRS, Orlando, Florida
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - UIC Project WISH CRS, Chicago, Illinois
  - VRC Clinical Trials Core CRS, Bethesda, Maryland
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Case Clinical Research Site, Cleveland, Ohio
  - Penn Prevention CRS, Philadelphia, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - University of Texas Southwestern CRS, Dallas, Texas
  - Baylor Vaccine Research Center CRS, Houston, Texas
  - Care-Id Crs, Annandale, Virginia
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Background] Lu S. Immunogenicity of DNA vaccines in humans: it takes two to tango. Hum Vaccin. 2008 Nov-Dec;4(6):449-52. doi: 10.4161/hv.4.6.6179. Epub 2008 Nov 28. PMID 18443427
- [Background] Patterson S, Papagatsias T, Benlahrech A. Use of adenovirus in vaccines for HIV. Handb Exp Pharmacol. 2009;(188):275-93. doi: 10.1007/978-3-540-71029-5_13. PMID 19031031
- [Result] Benmira S, Bhattacharya V, Schmid ML. An effective HIV vaccine: A combination of humoral and cellular immunity? Curr HIV Res. 2010 Sep;8(6):441-9. doi: 10.2174/157016210793499286. PMID 20636279
- [Derived] Hammer SM, Sobieszczyk ME, Janes H, Karuna ST, Mulligan MJ, Grove D, Koblin BA, Buchbinder SP, Keefer MC, Tomaras GD, Frahm N, Hural J, Anude C, Graham BS, Enama ME, Adams E, DeJesus E, Novak RM, Frank I, Bentley C, Ramirez S, Fu R, Koup RA, Mascola JR, Nabel GJ, Montefiori DC, Kublin J, McElrath MJ, Corey L, Gilbert PB; HVTN 505 Study Team. Efficacy trial of a DNA/rAd5 HIV-1 preventive vaccine. N Engl J Med. 2013 Nov 28;369(22):2083-92. doi: 10.1056/NEJMoa1310566. Epub 2013 Oct 7. PMID 24099601

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine: Participants will receive a recombinant DNA plasmid vaccine injection at study entry and on Days 28 and 56, followed by a recombinant adenoviral serotype vector vaccine injection on Day 168. As of April 2013, all vaccinations in this study have been stopped.
  DNA plasmid vaccine: 4-mg injection administered as 1 mL intramuscularly (IM) via Biojector® in either deltoid
  Recombinant adenoviral serotype 5 (rAD5) vector vaccine: 1 x 10^10 particle units (PU) administered as 1mL IM by needle and syringe in either deltoid
- Placebo: Participants will receive a recombinant DNA plasmid vaccine placebo injection at study entry and on Days 28 and 56, followed by a recombinant adenoviral serotype vector vaccine placebo injection on Day 168. As of April 2013, all vaccinations in this study have been stopped.
  DNA vaccine placebo: 1 mL IM via Biojector® in either deltoid
  HIV-1 recombinant adenovirus vaccine placebo: 1 mL administered IM by needle and syringe in either deltoid
Period: Overall Study
Arm/Group | Vaccine | Placebo
Started (Enrollment is defined as receiving the first vaccination.) | 1253 | 1251
Modified Intent-to-Treat Population (Participants excluded from MITT if HIV-1 positive at first vaccination (retrospective testing)) | 1251 | 1245
Completed (Completed if attended all visits. Note dropout endpoint does NOT include all visits.) | 629 | 564
Not Completed | 624 | 687
Not completed — Death | 1 | 11
Not completed — Lost to Follow-up | 314 | 315
Not completed — Withdrawal by Subject | 45 | 65
Not completed — Physician Decision | 0 | 1
Not completed — Participant relocated | 78 | 107
Not completed — Participant unable to adhere | 27 | 42
Not completed — Other; N=245 due to early study closure | 154 | 139
Not completed — HIV infection | 5 | 7

BASELINE CHARACTERISTICS:
Population: All Enrolled Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine | Placebo | Total
Number analyzed (Participants) | 1253 | 1251 | 2504
Age, Continuous [Median (Full Range); unit: years] | 29 [18 to 50] | 30 [18 to 50] | 29 [18 to 50]
Age, Customized [Count of Participants; unit: Participants]
  18-20 years | 105 | 108 | 213
  21-30 years | 585 | 569 | 1154
  31-40 years | 299 | 299 | 598
  41-50 years | 264 | 275 | 539
Sex/Gender, Customized [Count of Participants; unit: Participants] — Self-reported gender identity
  Participants
    Male | 1231 | 1229 | 2460
    Female | 4 | 4 | 8
    Transgender Male | 1 | 1 | 2
    Transgender Female | 13 | 15 | 28
    Other | 4 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1253 | 1251 | 2504
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 125 | 94 | 219
  Not Hispanic or Latino | 1128 | 1157 | 2285
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 10 | 13
  Asian | 13 | 20 | 33
  Native Hawaiian or Other Pacific Islander | 4 | 6 | 10
  Black or African American | 222 | 204 | 426
  White | 939 | 944 | 1883
  More than one race | 45 | 46 | 91
  Unknown or Not Reported | 27 | 21 | 48
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  <18.5 kg/m^2 | 22 | 16 | 38
  18.5-24.9 kg/m^2 | 550 | 586 | 1136
  25.0-29.9 kg/m^2 | 391 | 381 | 772
  30.0-34.9 kg/m^2 | 189 | 167 | 356
  35-39.9 kg/m^2 | 64 | 59 | 123
  >=40 kg/m^2 | 36 | 41 | 77
  Missing/Unknown | 1 | 1 | 2
Number of male sexual partners within 3 months prior to screening assessment [Count of Participants; unit: Participants]
  0 | 59 | 64 | 123
  1 | 256 | 243 | 499
  2 | 253 | 242 | 495
  3-4 | 349 | 367 | 716
  5 or more | 330 | 327 | 657
  Unknown | 6 | 8 | 14
Number of male sexual partners within 3 months prior to screening assessment [Median (Full Range); unit: partners] — Self-reported at screening
  partners | 3 [0 to 125] | 3 [0 to 70] | 3 [0 to 125]
Any unprotected receptive anal sex with a partner within 3 months prior to screening assessment [Count of Participants; unit: Participants] — Self-reported at screening
  Participants | 589 | 573 | 1162

OUTCOME MEASURES:

1. Primary Outcome: Participant Dropout Through Month 48
Description: For participants remaining uninfected, dropout is assessed only for primary follow-up, i.e. clinic visits. Protocol versions 4 and earlier included 24 months of primary follow-up, and versions 5 and later included 48 months. Participants may terminate early after completing primary follow-up, and participants who were found to be HIV-1 infected are analyzed as non-dropouts, so the number of dropouts and number of early terminations need not match.
Time Frame: Enrollment through Month 48 visit
Population: MITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1251 | 1245
Participants | 340 | 436
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Cox proportional hazards model to assess the association between treatment assignment and dropout; Test type: Other — Score test; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.63 to 0.84] — HR is vaccine / placebo

2. Primary Outcome: Participant Dropout Prior to Unblinding
Description: The trial was unblinded on April 23, 2013, and the protocol was in version 4 at the time.
  For participants remaining uninfected, dropout is assessed only for primary follow-up, i.e. clinic visits. Protocol versions 4 and earlier included 24 months of primary follow-up, and versions 5 and later included 48 months. Participants may terminate early after completing primary follow-up, and participants who were found to be HIV-1 infected are analyzed as non-dropouts, so the number of dropouts and number of early terminations need not match.
Time Frame: Enrollment until the date of dropout, through April 22, 2013 (up to Month 24 visit)
Population: MITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1251 | 1245
Participants | 99 | 127
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Cox PH model to assess the association between treatment assignment and dropout; Test type: Other; p = 0.05, Regression, Cox — Score test; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.59 to 1] — HR is vaccine / placebo

3. Primary Outcome: Participant Dropout After Unblinding
Description: as for outcome 2
Time Frame: April 23, 2013 through trial closure (up to Month 48 visit)
Population: MITT population participants who were HIV-uninfected and on-study as of April 23, 2013
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1036 | 999
Participants | 241 | 309
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Assess the association between treatment assignment and dropout; Test type: Other; p < 0.001, Regression, Cox — Score test; Cox Proportional Hazard = 0.71, 95% CI 2-sided [0.60 to 0.84] — HR is vaccine / placebo

4. Primary Outcome: HIV-1 Infections Diagnosed After Day 0 Including All Available Follow-up Through the Maximum Month 48 Visit
Description: For time-to-event analysis, an event is defined as HIV-1 infection and participants are censored if they dropped out early or completed the trial. HIV-1 diagnosis date is defined as the date of the earliest specimen collection yielding a positive HIV test. Participants remaining uninfected were censored at the latest specimen collection with a negative HIV-1 test.
Time Frame: Enrollment through Month 48 visit
Population: Modified Intent-to-Treat Cohort
Measure: Number; unit: participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1251 | 1245
participants | 75 | 68
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.903, Regression, Cox — Score test; Adjusted for age, behavioral risk score, square of behavioral risk score, race, and BMI; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.73 to 1.42] — HR is vaccine / placebo

5. Primary Outcome: HIV-1 Infections Diagnosed After Day 0 Through the Month 24 Visit
Description: For time-to-event analysis, an event is defined as HIV-1 infection and participants remaining uninfected through the month 24 visit were censored. HIV-1 diagnosis date is defined as the date of the earliest specimen collection at or prior to month 24 which yielded a positive HIV test. Participants remaining uninfected through the month 24 visit were censored at the latest specimen collection with a negative HIV-1 test at or prior to the month 24 visit.
Time Frame: Enrollment through Month 24 visit
Population: Modified Intent-to-Treat Cohort
Measure: Number; unit: participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1251 | 1245
participants | 49 | 46
Statistical Analysis 1: Comparison: Vaccine vs Placebo; Test type: Other; p = 0.783, Regression, Cox — Adjusted for ave, behavioral risk score, square of behavioral risk score, and BMI; Score test; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.71 to 1.58] — HR is vaccine / placebo

6. Primary Outcome: Number of Participants Experiencing Local Reactogenicity: Pain and/or Tenderness
Description: For each sign or symptom, we define the maximum observed grade for each participant over all vaccinations and post-vaccination assessments. Local and systemic signs and symptoms are assessed and graded based on The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December, 2004 (Clarification dated August 2009). Local reactogenicity parameters are pain, tenderness, erythema, and induration. We present the maximum grade for pain and/or tenderness, and erythema and/or induration.
Time Frame: Through 3 days post each study vaccination, and to resolution for events present at the third day post vaccination
Population: All Enrolled Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1253 | 1251
Participants
  None | 138 | 415
  Mild | 723 | 744
  Moderate | 370 | 90
  Severe | 22 | 2
  Potentially life-threatening | 0 | 0

7. Primary Outcome: Number of Participants Experiencing Local Reactogenicity: Erythema and/or Induration
Description: as for outcome 6
Time Frame: Through 3 days post each study vaccination, and to resolution for events present at the third day post vaccination
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1253 | 1251
Participants
  None | 717 | 980
  >0 to 25 square cm | 498 | 268
  >25 to 81 square cm (grade 1) | 15 | 2
  >9 cm any diameter (grade 2) | 6 | 0
  >81 square cm (grade 2) | 17 | 1

8. Primary Outcome: Number of Participants Experiencing Systemic Reactogenicity
Description: For each sign or symptom, we define the maximum observed grade for each participant over all vaccinations and post-vaccination assessments. Local and systemic signs and symptoms are assessed and graded based on The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December, 2004 (Clarification dated August 2009). Systemic reactogenicity parameters are malaise/fatigue, myalgia, headache, nausea, vomiting, chills, and arthralgia. We present the maximum grade calculated over these parameters.
Time Frame: Through 3 days post each study vaccination, and to resolution for events present at the third day post vaccination
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine | Placebo
Number analyzed (Participants) | 1253 | 1251
Participants
  None | 563 | 667
  Mild | 408 | 406
  Moderate | 240 | 169
  Severe | 42 | 9
  Potentially life-threatening | 0 | 0

ADVERSE EVENTS:
Time Frame: Reporting of all AEs occurred during 2 periods for each participant: 1) from enrollment through 28 days after the third vaccination, and 2) from the fourth vaccination through 28 days after the fourth vaccination. Between and after these time periods, only SAEs, new chronic conditions requiring medical intervention of more than 30 days, and newly diagnosed/treated STIs were reported. Events requiring expedited reporting (protocol section 12.3) were reported through the study, up to 60 months.
Arm/Group | Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/1253 | 11/1251
Serious Adverse Events (participants affected / at risk) | 77/1253 | 95/1251
Other Adverse Events (participants affected / at risk) | 833/1253 | 828/1251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=1253) | Placebo (N=1251)
Any event in SOC (Blood and lymphatic system disorders) | 0 | 1
Anaemias NEC (Blood and lymphatic system disorders) | 0 | 1
Any event in SOC (Cardiac disorders) | 1 | 6
Ischaemic coronary artery disorders (Cardiac disorders) | 1 | 2
Coronary artery disorders NEC (Cardiac disorders) | 0 | 1
Heart failures NEC (Cardiac disorders) | 0 | 1
Supraventricular arrhythmias (Cardiac disorders) | 0 | 1
Ventricular arrhythmias and cardiac arrest (Cardiac disorders) | 0 | 1
Any event in SOC (Congenital, familial and genetic disorders) | 0 | 1
Haemoglobinopathies congenital (Congenital, familial and genetic disorders) | 0 | 1
Any event in SOC (Gastrointestinal disorders) | 2 | 15
Colitis (excl infective) (Gastrointestinal disorders) | 1 | 3
Acute and chronic pancreatitis (Gastrointestinal disorders) | 1 | 1
Duodenal ulcers and perforation (Gastrointestinal disorders) | 0 | 2
Intestinal ulcers and perforation NEC (Gastrointestinal disorders) | 0 | 2
Abdominal hernias NEC (Gastrointestinal disorders) | 0 | 1
Gastric ulcers and perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal atonic and hypomotility disorders NEC (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders NEC (Gastrointestinal disorders) | 0 | 1
Gastrointestinal stenosis and obstruction NEC (Gastrointestinal disorders) | 0 | 1
Non-site specific gastrointestinal haemorrhages (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcers and perforation (Gastrointestinal disorders) | 0 | 1
Rectal inflammations NEC (Gastrointestinal disorders) | 0 | 1
Any event in SOC (General disorders) | 2 | 5
Pain and discomfort NEC (General disorders) | 1 | 3
Death and sudden death (General disorders) | 0 | 2
Withdrawal and rebound effects (General disorders) | 1 | 0
Any event in SOC (Immune system disorders) | 1 | 1
Acute and chronic sarcoidosis (Immune system disorders) | 0 | 1
Allergies to foods, food additives, drugs and other chemicals (Immune system disorders) | 1 | 0
Any event in SOC (Infections and infestations) | 25 | 26
Abdominal and gastrointestinal infections (Infections and infestations) | 8 | 11
Bacterial infections NEC (Infections and infestations) | 5 | 4
Infections NEC (Infections and infestations) | 2 | 3
Lower respiratory tract and lung infections (Infections and infestations) | 3 | 1
Upper respiratory tract infections (Infections and infestations) | 1 | 2
Clostridia infections (Infections and infestations) | 2 | 0
Sepsis, bacteraemia, viraemia and fungaemia NEC (Infections and infestations) | 1 | 1
Skin structures and soft tissue infections (Infections and infestations) | 1 | 1
Staphylococcal infections (Infections and infestations) | 2 | 0
Streptococcal infections (Infections and infestations) | 1 | 1
Bone and joint infections (Infections and infestations) | 1 | 0
Borrelial infections (Infections and infestations) | 1 | 0
Breast infections (Infections and infestations) | 0 | 1
Herpes viral infections (Infections and infestations) | 1 | 0
Infectious disorders carrier (Infections and infestations) | 1 | 0
Urinary tract infections (Infections and infestations) | 1 | 0
Viral infections NEC (Infections and infestations) | 0 | 1
Any event in SOC (Injury, poisoning and procedural complications) | 15 | 15
Limb fractures and dislocations (Injury, poisoning and procedural complications) | 4 | 2
Skull fractures, facial bone fractures and dislocations (Injury, poisoning and procedural complications) | 2 | 3
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 2 | 2
Overdoses NEC (Injury, poisoning and procedural complications) | 1 | 2
Poisoning and toxicity (Injury, poisoning and procedural complications) | 1 | 1
Site specific injuries NEC (Injury, poisoning and procedural complications) | 2 | 0
Skin injuries NEC (Injury, poisoning and procedural complications) | 1 | 1
Spinal fractures and dislocations (Injury, poisoning and procedural complications) | 0 | 2
Abdominal injuries NEC (Injury, poisoning and procedural complications) | 0 | 1
Cardiac and vascular procedural complications (Injury, poisoning and procedural complications) | 0 | 1
Cardiovascular injuries (Injury, poisoning and procedural complications) | 1 | 0
Cerebral injuries NEC (Injury, poisoning and procedural complications) | 1 | 0
Muscle, tendon and ligament injuries (Injury, poisoning and procedural complications) | 0 | 1
Pathways and sources of exposure (Injury, poisoning and procedural complications) | 0 | 1
Thermal burns (Injury, poisoning and procedural complications) | 1 | 0
Any event in SOC (Investigations) | 1 | 1
Liver function analyses (Investigations) | 0 | 1
Metabolism tests NEC (Investigations) | 1 | 0
Any event in SOC (Metabolism and nutrition disorders) | 1 | 0
Potassium imbalance (Metabolism and nutrition disorders) | 1 | 0
Any event in SOC (Musculoskeletal and connective tissue disorders) | 1 | 3
Bursal disorders (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorders NEC (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness conditions (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathies (Musculoskeletal and connective tissue disorders) | 0 | 1
Any event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Prostatic neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colorectal neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemias acute lymphocytic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testicular neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasms malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Any event in SOC (Nervous system disorders) | 7 | 2
Seizures and seizure disorders NEC (Nervous system disorders) | 3 | 0
Central nervous system haemorrhages and cerebrovascular accidents (Nervous system disorders) | 0 | 1
Encephalopathies NEC (Nervous system disorders) | 0 | 1
Mononeuropathies (Nervous system disorders) | 1 | 0
Neurological signs and symptoms NEC (Nervous system disorders) | 1 | 0
Optic nerve disorders NEC (Nervous system disorders) | 1 | 0
Transient cerebrovascular events (Nervous system disorders) | 1 | 0
Any event in SOC (Product Issues) | 0 | 1
Device malfunction events NEC (Product Issues) | 0 | 1
Any event in SOC (Psychiatric disorders) | 23 | 22
Suicidal and self-injurious behaviour (Psychiatric disorders) | 13 | 11
Depressive disorders (Psychiatric disorders) | 4 | 3
Substance related and addictive disorders (Psychiatric disorders) | 5 | 2
Bipolar disorders (Psychiatric disorders) | 0 | 3
Anxiety symptoms (Psychiatric disorders) | 1 | 1
Psychotic disorder NEC (Psychiatric disorders) | 0 | 2
Confusion and disorientation (Psychiatric disorders) | 1 | 0
Mental disorders NEC (Psychiatric disorders) | 1 | 0
Schizoaffective and schizophreniform disorders (Psychiatric disorders) | 1 | 0
Schizophrenia NEC (Psychiatric disorders) | 0 | 1
Somatic symptom disorders (Psychiatric disorders) | 1 | 0
Any event in SOC (Renal and urinary disorders) | 1 | 1
Renal failure and impairment (Renal and urinary disorders) | 1 | 0
Renal lithiasis (Renal and urinary disorders) | 0 | 1
Any event in SOC (Reproductive system and breast disorders) | 1 | 0
Testicular and epididymal disorders NEC (Reproductive system and breast disorders) | 1 | 0
Any event in SOC (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary thrombotic and embolic conditions (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax and pleural effusions NEC (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Any event in SOC (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue ulcerations (Skin and subcutaneous tissue disorders) | 1 | 0
Any event in SOC (Vascular disorders) | 4 | 1
Peripheral embolism and thrombosis (Vascular disorders) | 2 | 0
Non-site specific necrosis and vascular insufficiency NEC (Vascular disorders) | 0 | 1
Vascular hypertensive disorders NEC (Vascular disorders) | 1 | 0
Vascular hypotensive disorders (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine (N=1253) | Placebo (N=1251)
Any event in SOC (Blood and lymphatic system disorders) | 22 | 17
Lymphatic system disorders NEC (Blood and lymphatic system disorders) | 20 | 15
Anaemias NEC (Blood and lymphatic system disorders) | 2 | 0
Leukocytoses NEC (Blood and lymphatic system disorders) | 0 | 1
Red blood cell abnormal findings NEC (Blood and lymphatic system disorders) | 0 | 1
Spleen disorders (Blood and lymphatic system disorders) | 1 | 0
Any event in SOC (Cardiac disorders) | 2 | 5
Supraventricular arrhythmias (Cardiac disorders) | 1 | 2
Cardiac signs and symptoms NEC (Cardiac disorders) | 0 | 2
Rate and rhythm disorders NEC (Cardiac disorders) | 1 | 1
Any event in SOC (Congenital, familial and genetic disorders) | 1 | 1
Male reproductive tract disorders congenital (Congenital, familial and genetic disorders) | 1 | 1
Any event in SOC (Ear and labyrinth disorders) | 10 | 7
Ear disorders NEC (Ear and labyrinth disorders) | 3 | 5
Inner ear signs and symptoms (Ear and labyrinth disorders) | 3 | 1
External ear disorders NEC (Ear and labyrinth disorders) | 1 | 2
Middle ear disorders NEC (Ear and labyrinth disorders) | 2 | 0
Eustachian tube disorders (Ear and labyrinth disorders) | 1 | 0
Hearing losses (Ear and labyrinth disorders) | 0 | 1
Tympanic membrane disorders (excl infections) (Ear and labyrinth disorders) | 1 | 0
Any event in SOC (Endocrine disorders) | 8 | 2
Thyroid hypofunction disorders (Endocrine disorders) | 4 | 2
Endocrine abnormalities of gonadal function NEC (Endocrine disorders) | 2 | 0
Male gonadal function disorders (Endocrine disorders) | 1 | 0
Thyroid hyperfunction disorders (Endocrine disorders) | 1 | 0
Any event in SOC (Eye disorders) | 17 | 11
Lid, lash and lacrimal infections, irritations and inflammations (Eye disorders) | 4 | 1
Ocular disorders NEC (Eye disorders) | 2 | 2
Conjunctival and corneal bleeding and vascular disorders (Eye disorders) | 2 | 1
Ocular sensation disorders (Eye disorders) | 0 | 3
Visual disorders NEC (Eye disorders) | 3 | 0
Conjunctival infections, irritations and inflammations (Eye disorders) | 1 | 1
Eyelid movement disorders (Eye disorders) | 1 | 1
Lacrimation disorders (Eye disorders) | 2 | 0
Ocular infections, inflammations and associated manifestations (Eye disorders) | 1 | 1
Blindness (excl colour blindness) (Eye disorders) | 0 | 1
Glaucomas (excl congenital) (Eye disorders) | 1 | 0
Refractive and accommodative disorders (Eye disorders) | 1 | 0
Retinal, choroid and vitreous infections and inflammations (Eye disorders) | 0 | 1
Any event in SOC (Gastrointestinal disorders) | 149 | 146
Diarrhoea (excl infective) (Gastrointestinal disorders) | 53 | 53
Nausea and vomiting symptoms (Gastrointestinal disorders) | 28 | 21
Gastrointestinal and abdominal pains (excl oral and throat) (Gastrointestinal disorders) | 22 | 13
Stomatitis and ulceration (Gastrointestinal disorders) | 11 | 6
Gastrointestinal atonic and hypomotility disorders NEC (Gastrointestinal disorders) | 6 | 9
Haemorrhoids and gastrointestinal varices (excl oesophageal) (Gastrointestinal disorders) | 5 | 9
Anal and rectal disorders NEC (Gastrointestinal disorders) | 5 | 8
Gastrointestinal signs and symptoms NEC (Gastrointestinal disorders) | 7 | 6
Gastrointestinal disorders NEC (Gastrointestinal disorders) | 7 | 4
Dental pain and sensation disorders (Gastrointestinal disorders) | 6 | 4
Dyspeptic signs and symptoms (Gastrointestinal disorders) | 1 | 6
Intestinal haemorrhages (Gastrointestinal disorders) | 2 | 5
Gastritis (excl infective) (Gastrointestinal disorders) | 3 | 3
Colitis (excl infective) (Gastrointestinal disorders) | 0 | 4
Non-site specific gastrointestinal haemorrhages (Gastrointestinal disorders) | 2 | 2
Abdominal hernias NEC (Gastrointestinal disorders) | 2 | 1
Anal and rectal signs and symptoms (Gastrointestinal disorders) | 2 | 1
Dental and periodontal infections and inflammations (Gastrointestinal disorders) | 2 | 1
Diaphragmatic hernias (Gastrointestinal disorders) | 2 | 1
Flatulence, bloating and distension (Gastrointestinal disorders) | 1 | 2
Gingival disorders NEC (Gastrointestinal disorders) | 2 | 1
Gingival haemorrhages (Gastrointestinal disorders) | 2 | 1
Oesophageal ulcers and perforation (Gastrointestinal disorders) | 2 | 1
Tongue disorders (Gastrointestinal disorders) | 3 | 0
Tongue signs and symptoms (Gastrointestinal disorders) | 1 | 2
Benign neoplasms gastrointestinal (excl oral cavity) (Gastrointestinal disorders) | 0 | 2
Gastrointestinal inflammatory disorders NEC (Gastrointestinal disorders) | 2 | 0
Oral dryness and saliva altered (Gastrointestinal disorders) | 1 | 1
Abdominal findings abnormal (Gastrointestinal disorders) | 0 | 1
Anal and rectal pains (Gastrointestinal disorders) | 0 | 1
Dental disorders NEC (Gastrointestinal disorders) | 1 | 0
Faecal abnormalities NEC (Gastrointestinal disorders) | 0 | 1
Gastrointestinal dyskinetic disorders (Gastrointestinal disorders) | 0 | 1
Gastrointestinal fistulae (Gastrointestinal disorders) | 0 | 1
Inguinal hernias (Gastrointestinal disorders) | 0 | 1
Oral soft tissue pain and paraesthesia (Gastrointestinal disorders) | 0 | 1
Peptic ulcers and perforation (Gastrointestinal disorders) | 1 | 0
Rectal inflammations NEC (Gastrointestinal disorders) | 0 | 1
Any event in SOC (General disorders) | 138 | 104
Injection site reactions (General disorders) | 65 | 33
Asthenic conditions (General disorders) | 41 | 27
Febrile disorders (General disorders) | 17 | 15
Feelings and sensations NEC (General disorders) | 10 | 9
General signs and symptoms NEC (General disorders) | 6 | 10
Pain and discomfort NEC (General disorders) | 6 | 5
Administration site reactions NEC (General disorders) | 3 | 6
Oedema NEC (General disorders) | 2 | 5
Therapeutic and nontherapeutic responses (General disorders) | 2 | 4
Vaccination site reactions (General disorders) | 5 | 1
Mass conditions NEC (General disorders) | 0 | 3
Withdrawal and rebound effects (General disorders) | 2 | 1
Inflammations (General disorders) | 1 | 0
Any event in SOC (Hepatobiliary disorders) | 3 | 3
Hepatocellular damage and hepatitis NEC (Hepatobiliary disorders) | 2 | 1
Cholecystitis and cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholestasis and jaundice (Hepatobiliary disorders) | 0 | 1
Hepatobiliary signs and symptoms (Hepatobiliary disorders) | 1 | 0
Any event in SOC (Immune system disorders) | 25 | 14
Atopic disorders (Immune system disorders) | 10 | 7
Allergies to foods, food additives, drugs and other chemicals (Immune system disorders) | 9 | 5
Allergic conditions NEC (Immune system disorders) | 6 | 1
Anaphylactic and anaphylactoid responses (Immune system disorders) | 0 | 1
Any event in SOC (Infections and infestations) | 531 | 549
Upper respiratory tract infections (Infections and infestations) | 275 | 254
Neisseria infections (Infections and infestations) | 79 | 83
Viral infections NEC (Infections and infestations) | 75 | 72
Chlamydial infections (Infections and infestations) | 72 | 72
Treponema infections (Infections and infestations) | 32 | 41
Abdominal and gastrointestinal infections (Infections and infestations) | 37 | 29
Herpes viral infections (Infections and infestations) | 31 | 30
Streptococcal infections (Infections and infestations) | 22 | 31
Urinary tract infections (Infections and infestations) | 20 | 24
Lower respiratory tract and lung infections (Infections and infestations) | 16 | 14
Papilloma viral infections (Infections and infestations) | 12 | 17
Bacterial infections NEC (Infections and infestations) | 15 | 11
Eye and eyelid infections (Infections and infestations) | 9 | 17
Skin structures and soft tissue infections (Infections and infestations) | 11 | 14
Dental and oral soft tissue infections (Infections and infestations) | 9 | 14
Ectoparasitic infestations (Infections and infestations) | 8 | 15
Ear infections (Infections and infestations) | 8 | 10
Staphylococcal infections (Infections and infestations) | 10 | 5
Tinea infections (Infections and infestations) | 6 | 8
Influenza viral infections (Infections and infestations) | 5 | 5
Infections NEC (Infections and infestations) | 5 | 4
Male reproductive tract infections (Infections and infestations) | 3 | 5
Fungal infections NEC (Infections and infestations) | 5 | 1
Hepatitis viral infections (Infections and infestations) | 1 | 4
Candida infections (Infections and infestations) | 1 | 2
Molluscum contagiosum viral infections (Infections and infestations) | 1 | 2
Epstein-Barr viral infections (Infections and infestations) | 1 | 1
Giardia infections (Infections and infestations) | 1 | 1
Tuberculous infections (Infections and infestations) | 0 | 2
Amoebic infections (Infections and infestations) | 1 | 0
Bone and joint infections (Infections and infestations) | 0 | 1
Caliciviral infections (Infections and infestations) | 1 | 0
Clostridia infections (Infections and infestations) | 0 | 1
Coxsackie viral infections (Infections and infestations) | 1 | 0
Cytomegaloviral infections (Infections and infestations) | 1 | 0
Escherichia infections (Infections and infestations) | 0 | 1
Haemophilus infections (Infections and infestations) | 0 | 1
Helicobacter infections (Infections and infestations) | 1 | 0
Nematode infections (Infections and infestations) | 0 | 1
Any event in SOC (Injury, poisoning and procedural complications) | 108 | 101
Skin injuries NEC (Injury, poisoning and procedural complications) | 28 | 20
Muscle, tendon and ligament injuries (Injury, poisoning and procedural complications) | 24 | 23
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 13 | 9
Non-site specific procedural complications (Injury, poisoning and procedural complications) | 12 | 8
Limb fractures and dislocations (Injury, poisoning and procedural complications) | 9 | 10
Site specific injuries NEC (Injury, poisoning and procedural complications) | 8 | 8
Neurological and psychiatric procedural complications (Injury, poisoning and procedural complications) | 10 | 3
Bone and joint injuries NEC (Injury, poisoning and procedural complications) | 4 | 5
Thermal burns (Injury, poisoning and procedural complications) | 2 | 7
Exposures to agents or circumstances NEC (Injury, poisoning and procedural complications) | 4 | 2
Radiation injuries (Injury, poisoning and procedural complications) | 3 | 3
Cerebral injuries NEC (Injury, poisoning and procedural complications) | 3 | 2
Fractures and dislocations NEC (Injury, poisoning and procedural complications) | 1 | 4
Eye injuries NEC (Injury, poisoning and procedural complications) | 2 | 1
Skull fractures, facial bone fractures and dislocations (Injury, poisoning and procedural complications) | 0 | 3
Thoracic cage fractures and dislocations (Injury, poisoning and procedural complications) | 1 | 2
Chest and lung injuries NEC (Injury, poisoning and procedural complications) | 2 | 0
Gastrointestinal and hepatobiliary procedural complications (Injury, poisoning and procedural complications) | 0 | 2
Ear injuries NEC (Injury, poisoning and procedural complications) | 0 | 1
Overdoses NEC (Injury, poisoning and procedural complications) | 1 | 0
Poisoning and toxicity (Injury, poisoning and procedural complications) | 1 | 0
Reproductive system and breast injuries (Injury, poisoning and procedural complications) | 0 | 1
Spinal fractures and dislocations (Injury, poisoning and procedural complications) | 0 | 1
Vaccination related complications (Injury, poisoning and procedural complications) | 1 | 0
Any event in SOC (Investigations) | 39 | 63
Vascular tests NEC (incl blood pressure) (Investigations) | 28 | 47
Reproductive hormone analyses (Investigations) | 3 | 7
Liver function analyses (Investigations) | 3 | 3
Red blood cell analyses (Investigations) | 2 | 2
Carbohydrate tolerance analyses (incl diabetes) (Investigations) | 2 | 1
Digestive enzymes (Investigations) | 2 | 0
Mineral and electrolyte analyses (Investigations) | 2 | 0
Platelet analyses (Investigations) | 0 | 2
Bacteria identification and serology (excl mycobacteria) (Investigations) | 0 | 1
Cardiac auscultatory investigations (Investigations) | 1 | 0
Coagulation and bleeding analyses (Investigations) | 1 | 0
Heart rate and pulse investigations (Investigations) | 1 | 0
Investigations NEC (Investigations) | 0 | 1
Musculoskeletal and soft tissue tests NEC (Investigations) | 1 | 0
Mycobacteria identification and serology (Investigations) | 0 | 1
Tissue enzyme analyses NEC (Investigations) | 1 | 0
White blood cell analyses (Investigations) | 0 | 1
Any event in SOC (Metabolism and nutrition disorders) | 27 | 20
Diabetes mellitus (incl subtypes) (Metabolism and nutrition disorders) | 7 | 3
Fat soluble vitamin deficiencies and disorders (Metabolism and nutrition disorders) | 3 | 5
Appetite disorders (Metabolism and nutrition disorders) | 5 | 1
Elevated cholesterol (Metabolism and nutrition disorders) | 2 | 3
Disorders of purine metabolism (Metabolism and nutrition disorders) | 3 | 0
General nutritional disorders NEC (Metabolism and nutrition disorders) | 2 | 1
Potassium imbalance (Metabolism and nutrition disorders) | 2 | 1
Fluid intake increased (Metabolism and nutrition disorders) | 2 | 0
Food malabsorption and intolerance syndromes (excl sugar intolerance) (Metabolism and nutrition disorders) | 1 | 1
Lipid metabolism and deposit disorders NEC (Metabolism and nutrition disorders) | 2 | 0
Water soluble vitamin deficiencies (Metabolism and nutrition disorders) | 1 | 1
Elevated triglycerides (Metabolism and nutrition disorders) | 0 | 1
Hyperlipidaemias NEC (Metabolism and nutrition disorders) | 0 | 1
Hypoglycaemic conditions NEC (Metabolism and nutrition disorders) | 0 | 1
Magnesium metabolism disorders (Metabolism and nutrition disorders) | 0 | 1
Protein metabolism disorders NEC (Metabolism and nutrition disorders) | 1 | 0
Sugar intolerance (excl glucose intolerance) (Metabolism and nutrition disorders) | 0 | 1
Total fluid volume decreased (Metabolism and nutrition disorders) | 0 | 1
Any event in SOC (Musculoskeletal and connective tissue disorders) | 97 | 107
Musculoskeletal and connective tissue pain and discomfort (Musculoskeletal and connective tissue disorders) | 47 | 49
Muscle pains (Musculoskeletal and connective tissue disorders) | 25 | 24
Joint related signs and symptoms (Musculoskeletal and connective tissue disorders) | 17 | 19
Muscle related signs and symptoms NEC (Musculoskeletal and connective tissue disorders) | 7 | 2
Tendon disorders (Musculoskeletal and connective tissue disorders) | 3 | 3
Bone related signs and symptoms (Musculoskeletal and connective tissue disorders) | 2 | 3
Arthropathies NEC (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone disorders NEC (Musculoskeletal and connective tissue disorders) | 1 | 2
Bursal disorders (Musculoskeletal and connective tissue disorders) | 1 | 2
Intervertebral disc disorders NEC (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle weakness conditions (Musculoskeletal and connective tissue disorders) | 0 | 3
Muscle tone abnormalities (Musculoskeletal and connective tissue disorders) | 0 | 2
Cartilage disorders (Musculoskeletal and connective tissue disorders) | 1 | 0
Extremity deformities (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint related disorders NEC (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue infections and inflammations NEC (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthropathies (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthropathies (Musculoskeletal and connective tissue disorders) | 1 | 0
Soft tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial disorders (Musculoskeletal and connective tissue disorders) | 1 | 0
Any event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 17
Skin neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 14
Lip and oral cavity neoplasms benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Skin neoplasms malignant and unspecified (excl melanoma) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Soft tissue neoplasms benign NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Nervous system neoplasms benign NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Reproductive neoplasms male benign NEC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Any event in SOC (Nervous system disorders) | 103 | 88
Headaches NEC (Nervous system disorders) | 39 | 41
Neurological signs and symptoms NEC (Nervous system disorders) | 30 | 22
Paraesthesias and dysaesthesias (Nervous system disorders) | 10 | 11
Migraine headaches (Nervous system disorders) | 8 | 2
Sensory abnormalities NEC (Nervous system disorders) | 8 | 1
Disturbances in consciousness NEC (Nervous system disorders) | 7 | 1
Mononeuropathies (Nervous system disorders) | 2 | 3
Peripheral neuropathies NEC (Nervous system disorders) | 4 | 1
Lumbar spinal cord and nerve root disorders (Nervous system disorders) | 2 | 1
Narcolepsy and hypersomnia (Nervous system disorders) | 1 | 1
Seizures and seizure disorders NEC (Nervous system disorders) | 1 | 1
Cervical spinal cord and nerve root disorders (Nervous system disorders) | 0 | 1
Coordination and balance disturbances (Nervous system disorders) | 0 | 1
Disturbances in sleep phase rhythm (Nervous system disorders) | 0 | 1
Facial cranial nerve disorders (Nervous system disorders) | 0 | 1
Memory loss (excl dementia) (Nervous system disorders) | 1 | 0
Mental impairment (excl dementia and memory loss) (Nervous system disorders) | 0 | 1
Neurologic visual problems NEC (Nervous system disorders) | 1 | 0
Sleep disturbances NEC (Nervous system disorders) | 1 | 0
Any event in SOC (Psychiatric disorders) | 72 | 65
Depressive disorders (Psychiatric disorders) | 25 | 22
Anxiety symptoms (Psychiatric disorders) | 20 | 17
Disturbances in initiating and maintaining sleep (Psychiatric disorders) | 8 | 12
Substance related and addictive disorders (Psychiatric disorders) | 9 | 4
Attention deficit and disruptive behaviour disorders (Psychiatric disorders) | 3 | 4
Anxiety disorders NEC (Psychiatric disorders) | 5 | 1
Bipolar disorders (Psychiatric disorders) | 2 | 3
Panic attacks and disorders (Psychiatric disorders) | 3 | 2
Sexual desire disorders (Psychiatric disorders) | 3 | 2
Stress disorders (Psychiatric disorders) | 2 | 1
Emotional and mood disturbances NEC (Psychiatric disorders) | 0 | 2
Schizophrenia NEC (Psychiatric disorders) | 2 | 0
Behaviour and socialisation disturbances (Psychiatric disorders) | 0 | 1
Fear symptoms and phobic disorders (incl social phobia) (Psychiatric disorders) | 0 | 1
Fluctuating mood symptoms (Psychiatric disorders) | 1 | 0
Mental disorders NEC (Psychiatric disorders) | 1 | 0
Mood alterations with depressive symptoms (Psychiatric disorders) | 1 | 0
Mood disorders NEC (Psychiatric disorders) | 0 | 1
Schizoaffective and schizophreniform disorders (Psychiatric disorders) | 1 | 0
Sleep disorders NEC (Psychiatric disorders) | 0 | 1
Somatic symptom disorders (Psychiatric disorders) | 1 | 0
Suicidal and self-injurious behaviour (Psychiatric disorders) | 0 | 1
Any event in SOC (Renal and urinary disorders) | 19 | 23
Bladder and urethral symptoms (Renal and urinary disorders) | 11 | 12
Renal lithiasis (Renal and urinary disorders) | 4 | 6
Urethral disorders NEC (Renal and urinary disorders) | 1 | 4
Urinary abnormalities (Renal and urinary disorders) | 1 | 2
Urinary tract signs and symptoms NEC (Renal and urinary disorders) | 2 | 1
Bladder neoplasms (Renal and urinary disorders) | 1 | 0
Any event in SOC (Reproductive system and breast disorders) | 27 | 26
Penile disorders NEC (excl erection and ejaculation) (Reproductive system and breast disorders) | 12 | 7
Reproductive tract signs and symptoms NEC (Reproductive system and breast disorders) | 5 | 4
Erection and ejaculation conditions and disorders (Reproductive system and breast disorders) | 1 | 5
Prostate and seminal vesicles infections and inflammations (Reproductive system and breast disorders) | 2 | 4
Reproductive tract disorders NEC (excl neoplasms) (Reproductive system and breast disorders) | 3 | 1
Testicular and epididymal disorders NEC (Reproductive system and breast disorders) | 3 | 1
Breast signs and symptoms (Reproductive system and breast disorders) | 0 | 2
Scrotal disorders NEC (Reproductive system and breast disorders) | 0 | 2
Breast disorders NEC (Reproductive system and breast disorders) | 1 | 0
Pelvic prolapse conditions (Reproductive system and breast disorders) | 0 | 1
Sexual function and fertility disorders NEC (Reproductive system and breast disorders) | 1 | 0
Spermatogenesis and semen disorders (Reproductive system and breast disorders) | 1 | 0
Testicular and epididymal neoplasms (Reproductive system and breast disorders) | 0 | 1
Any event in SOC (Respiratory, thoracic and mediastinal disorders) | 123 | 95
Upper respiratory tract signs and symptoms (Respiratory, thoracic and mediastinal disorders) | 49 | 44
Coughing and associated symptoms (Respiratory, thoracic and mediastinal disorders) | 34 | 24
Nasal congestion and inflammations (Respiratory, thoracic and mediastinal disorders) | 22 | 17
Paranasal sinus disorders (excl infections and neoplasms) (Respiratory, thoracic and mediastinal disorders) | 15 | 10
Bronchospasm and obstruction (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Pharyngeal disorders (excl infections and neoplasms) (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Breathing abnormalities (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Nasal disorders NEC (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Respiratory tract disorders NEC (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Laryngeal and adjacent sites disorders NEC (excl infections and neoplasms) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedemas (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failures (excl neonatal) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Any event in SOC (Skin and subcutaneous tissue disorders) | 112 | 86
Dermatitis and eczema (Skin and subcutaneous tissue disorders) | 29 | 17
Rashes, eruptions and exanthems NEC (Skin and subcutaneous tissue disorders) | 21 | 25
Apocrine and eccrine gland disorders (Skin and subcutaneous tissue disorders) | 17 | 11
Dermal and epidermal conditions NEC (Skin and subcutaneous tissue disorders) | 11 | 11
Pruritus NEC (Skin and subcutaneous tissue disorders) | 14 | 8
Erythemas (Skin and subcutaneous tissue disorders) | 7 | 2
Psoriatic conditions (Skin and subcutaneous tissue disorders) | 6 | 3
Acnes (Skin and subcutaneous tissue disorders) | 3 | 3
Angioedemas (Skin and subcutaneous tissue disorders) | 2 | 1
Bullous conditions (Skin and subcutaneous tissue disorders) | 2 | 1
Papulosquamous conditions (Skin and subcutaneous tissue disorders) | 1 | 2
Pilar disorders NEC (Skin and subcutaneous tissue disorders) | 1 | 1
Purpura and related conditions (Skin and subcutaneous tissue disorders) | 1 | 1
Skin and subcutaneous tissue ulcerations (Skin and subcutaneous tissue disorders) | 2 | 0
Skin cysts and polyps (Skin and subcutaneous tissue disorders) | 1 | 1
Skin preneoplastic conditions NEC (Skin and subcutaneous tissue disorders) | 2 | 0
Alopecias (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis ascribed to specific agent (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperkeratoses (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperpigmentation disorders (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity and photodermatosis conditions (Skin and subcutaneous tissue disorders) | 0 | 1
Rosaceas (Skin and subcutaneous tissue disorders) | 0 | 1
Any event in SOC (Social circumstances) | 0 | 1
Crime victims (Social circumstances) | 0 | 1
Any event in SOC (Vascular disorders) | 33 | 49
Vascular hypertensive disorders NEC (Vascular disorders) | 25 | 42
Peripheral vascular disorders NEC (Vascular disorders) | 5 | 4
Haemorrhages NEC (Vascular disorders) | 2 | 2
Lymphoedemas (Vascular disorders) | 1 | 0
Peripheral embolism and thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-07-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT00865566/Prot_000.pdf
  • Statistical Analysis Plan (2014-10-03): https://cdn.clinicaltrials.gov/large-docs/66/NCT00865566/SAP_001.pdf